CLINICAL TRIAL: NCT03570944
Title: Postoperative Outcomes Within an Enhanced Recovery After Surgery Protocol National Audit of Complications Following Elective Total Hip or Knee Replacement Within or Without an Enhanced Recovery After Surgery Protocol (POWER2)
Brief Title: Postoperative Outcomes Within an Enhanced Recovery After Surgery Protocol (POWER2)
Acronym: POWER2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grupo Español de Rehabilitación Multimodal (Other)
Responsible Party: Sponsor
Other Study IDs: RedGerm02
Record Dates: First submitted 2018-06-17; First posted 2018-06-27 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Lysine-tRNA Ligase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing elective HRS or KRS: Adult patients undergoing elective HRS or KNS
  Interventions: Procedure: HRS, KRS

INTERVENTIONS:
Procedure: HRS, KRS — Elective HRS or KNR in adult patients, with any ERAS compliance

SUMMARY:
Methods National audit of a 60-day prospective observational cohort in the that the pre-defined postoperative complications at 30 days of follow-up in adult patients electively undergoing hip replacement surgery (HRS) or knee replacement surgery (KRS) with or without a program of Enhanced Recovery (ERAS: Enhanced Recovery after Surgery) with any level of protocol compliance (0-100%)

Research Places Spanish Hospitals where these surgical interventions are performed usually

Objectives To determine the incidence of Postoperative Complications per patient and procedure, regardless of the degree of adherence to ERAS protocols and its impact on the Hospital Stay and on postoperative complications including 30-day mortality

Sample Size For an alpha error of 5% (95% confidence and an accuracy of 3% and estimating a number of patients with complications of 50%, the calculation of sample size yields 3012 patients, although the final sample size may be smaller depending on the proportion of complications detected.

Inclusion criteria Patients over 18 undergoing elective HRS or KRS PTC regardless of its affiliation to a ERAS program and the level of compliance with protocol (from 0-100%)

Statistical analysis Continuous variables will be described as mean and standard deviation, if it is a normal distribution, or median and interquartile range, if they are not distributed normally. The comparisons of continuous variables are performed by one-way ANOVA or the Mann-Whitney test, depending on proceed A univariate analysis will be carried out to test the factors associated with postoperative complications, hospital stay and death in Hospital. Univariate analyzes and logistic regression models will be constructed Hierarchical multivariate to identify the factors associated in a independent with these results and to adjust the differences in the factors of confusion. The factors will be introduced in the models based on their relationship with the univariate result (p <0.05), the biological plausibility and the low rate of missing data.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 who undergoing HRS or KRS with or without an ERAS intensified recovery program with any level of protocol compliance (0-100%) Surgeries planned by inclusion criteria

  * Total elective knee replacement surgery(primary)
  * Total elective hip replacement surgery (primary)

Exclusion Criteria:

* Patients undergoing emergency surgery.

  * Partial prostheses
  * Replacement of prosthesis
  * Patients who decline to participate

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients
Sampling Method: Non-Probability Sample
Enrollment: 3012 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-28 (Estimated)

PRIMARY OUTCOMES:
30 day postoperative complications | 30 days
  Complications are defined according to Standards for definitions and use of outcomes for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions (1), the standardized list and definitions of the Knee Society (2) and Standardized List , Definitions, and the Stratification Developed by The Hip Society (3)

SECONDARY OUTCOMES:
Mortality | 30 day
  30 day mortality
Hospital Stay | 30 day
  Primary hospital stay after surgery

OTHER OUTCOMES:
ERAS overall compliance | 30 day
  ERAS compliance according to (4)

CONTACTS AND LOCATIONS:
Overall Officials: Ane Abad Motos, MD, Study Director — Infanta Leonor University Hospital
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Under request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years
Access Criteria: Mail to: power2@grupogerm.es
URL: http://www

REFERENCES:
- [Result] Jammer I, Wickboldt N, Sander M, Smith A, Schultz MJ, Pelosi P, Leva B, Rhodes A, Hoeft A, Walder B, Chew MS, Pearse RM; European Society of Anaesthesiology (ESA) and the European Society of Intensive Care Medicine (ESICM); European Society of Anaesthesiology; European Society of Intensive Care Medicine. Standards for definitions and use of outcome measures for clinical effectiveness research in perioperative medicine: European Perioperative Clinical Outcome (EPCO) definitions: a statement from the ESA-ESICM joint taskforce on perioperative outcome measures. Eur J Anaesthesiol. 2015 Feb;32(2):88-105. doi: 10.1097/EJA.0000000000000118. PMID 25058504
- [Result] Healy WL, Della Valle CJ, Iorio R, Berend KR, Cushner FD, Dalury DF, Lonner JH. Complications of total knee arthroplasty: standardized list and definitions of the Knee Society. Clin Orthop Relat Res. 2013 Jan;471(1):215-20. doi: 10.1007/s11999-012-2489-y. PMID 22810157
- [Result] Healy WL, Iorio R, Pellegrini VD, Della Valle CJ, Berend KR. Reply to the Letter to the Editor: Complications of Total Hip Arthroplasty: Standardized List, Definitions, and Stratification Developed by the Hip Society. Clin Orthop Relat Res. 2016 Jun;474(6):1528-9. doi: 10.1007/s11999-016-4804-5. Epub 2016 Apr 4. No abstract available. PMID 27043725
- [Result] Berend KR, Lombardi AV Jr, Mallory TH. Rapid recovery protocol for peri-operative care of total hip and total knee arthroplasty patients. Surg Technol Int. 2004;13:239-47. PMID 15744696
- [Derived] Ripolles-Melchor J, Abad-Motos A, Logrono-Egea M, Aldecoa C, Garcia-Erce JA, Jimenez-Lopez I, Cassinello-Ogea C, Marin-Pena O, Ferrando-Ortola C, de la Rica AS, Gomez-Rios MA, Sanchez-Martin R, Abad-Gurumeta A, Casans-Frances R, Mugarra-Llopis A, Varela-Duran M, Longas-Valien J, Ramiro-Ruiz A, Cuellar-Martinez AB, Ramirez-Rodriguez JM, Calvo-Vecino JM. Postoperative Outcomes Within Enhanced Recovery After Surgery Protocol in Elective Total Hip and Knee Arthroplasty. POWER.2 Study: Study Protocol for a Prospective, Multicentre, Observational Cohort Study. Turk J Anaesthesiol Reanim. 2019 Jun;47(3):179-186. doi: 10.5152/TJAR.2019.87523. Epub 2019 Jan 24. PMID 31183463